CLINICAL TRIAL: NCT02158065
Title: A 3-month Multicenter Randomized Trial to Evaluate the Efficacy of a Physical Activity Promotion Program on the Experience of Physical Activity in Patients With COPD (Mr PAPP)
Brief Title: Impact of "Telecoaching Program" on Physical Activity in Patients With COPD
Acronym: MrPAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University of Edinburgh (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); University Medical Center Groningen (Other); University of Athens (Other); University of Zurich (Other); Barcelona Institute for Global Health (Other)
Responsible Party: Principal Investigator, Thierry Troosters, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML9814
Record Dates: First submitted 2014-06-05; First posted 2014-06-06 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic obstructive pulmonary disease (COPD); physical activity; PROactive; telecoaching
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients will receive information (leaflet) and guidance on the benefits associated with increased physical activity in COPD patients and their health status
- Coaching program (Experimental): In addition to usual care, patients will receive the coaching program
  Interventions: Other: Coaching program

INTERVENTIONS:
Other: Coaching program — The coaching program consists of a (1) Step counter used as a coaching activity monitor to collect number of steps walked by the patients and (2) the Linkcare System, a mobile phone or tablet PC placed in the patient's home to collect data from the step counter. The system will set a daily activity goal for the patient based on achieved activity levels which will be measured by the step counter. Patients will also receive feedback, motivational and educational messages and direct calls from the coaching team at each institution.
  Arms: Coaching program

SUMMARY:
The purpose of this 3 month randomized intervention study is to investigate the additional effect of a physical activity telecoaching program on physical activity in patients with COPD, compared with usual care.

DETAILED DESCRIPTION:
In this 3 month, randomized (1:1 ratio), parallel-group, multicenter trial, patients in both groups (control and coaching) will receive information and guidance on the benefits associated with increased physical activity in COPD patients and their health status. Patients in both groups will use two PROactive monitors (ActiGraph® and DynaPort®) and a PDA to complete the PROactive questionnaire. In addition to above, the patients in the coaching group will receive daily coaching by a semiautomated system and coaching by the investigator during study visits.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Male and female patients ≥ 40 years of age
* Diagnosis of COPD (GOLD criteria: post bronchodilator FEV1/FVC< 70%)
* Current or ex-smokers with a smoking history equivalent to at least 10 pack years
* Patient should have at least 4 days of physical activity data recorded via PROactive monitors during 7 days prior to the baseline measurement

Exclusion Criteria:

* Orthopedic, neurological or other complaints that significantly impair normal biomechanical movement patterns, as judged by the investigator. Specifically if the patients' condition/ co-morbidities are such that physical activity cannot be increased, then they should not be enrolled
* Respiratory diseases other than COPD (e.g. asthma)
* Cognitive reading impairment and/or difficulties to manage electronic devices precluding interaction with the smartphone and PDA, as judged by the investigator
* Participating in or scheduled to start an outpatient rehabilitation program during the study. If the patient wishes to participate in pulmonary rehabilitation for any reason the patient can be enrolled in the study only at the end of rehabilitation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Daily number of steps | changes from baseline to 3 months
  The daily number of steps will be measured by the PROactive monitors (ActiGraph® and DynaPort®) at baseline (during the week prior to baseline visit) and at the end of the 3-month epoch (during the week prior to end visit).

SECONDARY OUTCOMES:
Time spent in at least moderate physical activity | changes from baseline to 3 months
  Time in at least moderate physical activity will be measured by the PROactive monitors (ActiGraph® and DynaPort®) at baseline (during the week prior to baseline visit) and at the end of the 3-month epoch (during the week prior to end visit).
Proportion of patients showing an increase of physical activity by >20% | changes from baseline to 3 months
  Physical activity will be measured by the PROactive monitors (ActiGraph® and DynaPort®) at baseline (during the week prior to baseline visit) and at the end of the 3-month epoch (during the week prior to end visit).
6-minute walking test | changes from baseline to 3 months
isometric Quadriceps force | changes from baseline to 3 months
COPD symptoms and health-related quality of life | changes form baseline to 3 months
  COPD symptoms and health-related quality of life will be measured by the CAT, CCQ, HADS and mMRC questionnaires

OTHER OUTCOMES:
daily and clinic visit version of PROactive instrument | changes from baseline to 3 months
Satisfaction with the telecoaching program | Information gathered after 3 months of intervention
  Questionnaire and qualitative interview about the patients' experience
Compliance with the telecoaching program | Information gathered after 3 months of intervention
  Compliance of wearing the step counter and performing the tasks of the smartphone interface

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Troosters, PT, PHD, Study Chair — KU Leuven; Mike Polkey, MD, PHD, Study Chair — Royal Brompton & Harefield NHS Foundation Trust; Judith Garcia-Aymerich, MD, PHD, Study Chair — Barcelona Institute for Global Health
Locations (6):
- KULeuven, Leuven, Belgium
- Thorax Research Foundation, Athens, Greece
- University Medical Center, Groningen, Netherlands
- University of Zurich, Zurich, Switzerland
- United Kingdom (2):
  - University of Edinburgh, Edinburgh
  - Royal Brompton Hospital, Imperial College, London

REFERENCES:
- [Derived] Loeckx M, Rabinovich RA, Demeyer H, Louvaris Z, Tanner R, Rubio N, Frei A, De Jong C, Gimeno-Santos E, Rodrigues FM, Buttery SC, Hopkinson NS, Busching G, Strassmann A, Serra I, Vogiatzis I, Garcia-Aymerich J, Polkey MI, Troosters T. Smartphone-Based Physical Activity Telecoaching in Chronic Obstructive Pulmonary Disease: Mixed-Methods Study on Patient Experiences and Lessons for Implementation. JMIR Mhealth Uhealth. 2018 Dec 21;6(12):e200. doi: 10.2196/mhealth.9774. PMID 30578215
- [Derived] Demeyer H, Louvaris Z, Frei A, Rabinovich RA, de Jong C, Gimeno-Santos E, Loeckx M, Buttery SC, Rubio N, Van der Molen T, Hopkinson NS, Vogiatzis I, Puhan MA, Garcia-Aymerich J, Polkey MI, Troosters T; Mr Papp PROactive study group and the PROactive consortium. Physical activity is increased by a 12-week semiautomated telecoaching programme in patients with COPD: a multicentre randomised controlled trial. Thorax. 2017 May;72(5):415-423. doi: 10.1136/thoraxjnl-2016-209026. Epub 2017 Jan 30. PMID 28137918